CLINICAL TRIAL: NCT05469685
Title: Efficacy and Safety of Vonoprazan- Amoxicillin Dual Therapy for Helicobacter Pylori Eradication : a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Dual Therapy for Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20220701-06
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; dual therapy; infection eradication; safety
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-day treatment group (Experimental): vonoprazan 20mg bid and amoxicillin 1000mg tid for 10 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- 14-day treatment group (Active Comparator): vonoprazan 20mg bid and amoxicillin 1000mg tid for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin

INTERVENTIONS:
Drug: Vonoprazan — Potassium-competitive acid blocker
Drug: Amoxicillin — Antibiotic for H. pylori eradication

SUMMARY:
The purpose of this study was to evaluate the Efficacy and Safety of Vonoprazan- amoxicillin dual therapy for Helicobacter Pylori eradication

DETAILED DESCRIPTION:
This study intends to select the patients with Hp infection in 11 tertiary hospitals across our country, and randomly give the two therapies to compare the eradication rate, compliance, the rate of adverse events, so as to provide some advices for the selection of appropriate eradication therapy, then collect an efficient, convenient and safe therapy for patients with H.pylori infection.

Before receiving the treatment plan, general information and relevant medical history of the subjects were collected through electronic questionnaires.The experimental data will be collected and recorded through follow-up by phone or WeChat during the experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 65 years; Sexes eligible for study: both;
2. patients who are diagnosed with Helicobacter pylori;
3. treatment-naive patients or patients who failed to eradicate Helicobacter pylori in the past but haven't undergone eradication therapy in the past six months;
4. voluntary to be involved in the study and written informed consent was obtained from all patients

Exclusion Criteria:

1. allergic reactions to the study drugs;
2. patients with peptic ulcer;
3. patients who underwent eradication therapy for Helicobacter pylori during the last six months;
4. patients who took antibiotics,bismuth agents,probiotics within four weeks prior to treatment and those who took H2 receptor antagonists,proton pump inhibitors(PPIs) or potassium competitive acid blockers within two weeks prior to treatment;
5. patients who are taking glucocorticoids, non-steroidal anti-inflammatory drugs or anticoagulants;
6. patients who have history of esophageal or gastric surgery;
7. pregnant or lactating women;
8. patients who have severe concurrent diseases such as hepatic,cardiovascular,respiratory,renal disorders or malignancies;
9. Alcohol abusers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | four to six weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by ¹³C-urea breath test four to six weeks after completion of the medication. The eradication rates will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
Adverse events | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types: dose-related, non-dose-related, dose-related and time-related, time-related, withdrawal, and failure of therapy.
Compliance Rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (10):
- China (10):
  - Affiliated Hospital of Integrated Traditional Chinese and Western Medicine, Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Changshu No.1 People's Hospital, Suzhou, Jiangsu
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Taixing People's Hospital, Taizhou, Jiangsu
  - Taizhou Fourth People's Hospital, Taizhou, Jiangsu
  - Wuxi People's Hospital Affiliated to Nanjing Medical University, Wuxi, Jiangsu
  - The First People's Hospital of Xuzhou, Xuzhou Municipal Hospital Affiliated to Xuzhou Medical University, Xuzhou, Jiangsu
  - Yancheng First Hospital,Affiliated Hospital of Nanjing University Medical School, Yancheng, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502
- [Background] Ford AC, Malfertheiner P, Giguere M, Santana J, Khan M, Moayyedi P. Adverse events with bismuth salts for Helicobacter pylori eradication: systematic review and meta-analysis. World J Gastroenterol. 2008 Dec 28;14(48):7361-70. doi: 10.3748/wjg.14.7361. PMID 19109870
- [Background] Rimbara E, Noguchi N, Kawai T, Sasatsu M. Mutations in penicillin-binding proteins 1, 2 and 3 are responsible for amoxicillin resistance in Helicobacter pylori. J Antimicrob Chemother. 2008 May;61(5):995-8. doi: 10.1093/jac/dkn051. Epub 2008 Feb 14. PMID 18276599
- [Background] Furuta T, Graham DY. Pharmacologic aspects of eradication therapy for Helicobacter pylori Infection. Gastroenterol Clin North Am. 2010 Sep;39(3):465-80. doi: 10.1016/j.gtc.2010.08.007. PMID 20951912
- [Background] Gao CP, Zhang D, Zhang T, Wang JX, Han SX, Graham DY, Lu H. PPI-amoxicillin dual therapy for Helicobacter pylori infection: An update based on a systematic review and meta-analysis. Helicobacter. 2020 Aug;25(4):e12692. doi: 10.1111/hel.12692. Epub 2020 Apr 20. PMID 32314468
- [Background] Berry V, Jennings K, Woodnutt G. Bactericidal and morphological effects of amoxicillin on Helicobacter pylori. Antimicrob Agents Chemother. 1995 Aug;39(8):1859-61. doi: 10.1128/AAC.39.8.1859. PMID 7486933
- [Derived] Dong Y, Duan Z, Liu M, Ding Y, Chen G, Wang R, Xu X, Ding L, Zhan Q, Pan C, Li H, Yang F, Dai X, Li X, Wu X, Peng P, Wang J, Hu K, Hu D, Jie Q, Zhang Z. Efficacy and cost-effectiveness analysis of 10-day versus 14-day eradication of Helicobacter pylori infection with vonoprazan amoxicillin: a prospective, multicenter, randomized controlled trial. Front Pharmacol. 2025 Mar 24;16:1543352. doi: 10.3389/fphar.2025.1543352. eCollection 2025. PMID 40196374